CLINICAL TRIAL: NCT00804609
Title: A Study to Evaluate the Effects of Epidural Lidocaine Administration on the Pharmacokinetic and Pharmacodynamic Profiles of DepoDur® (Morphine Sulfate Extended-release Injection) in Patients Undergoing Cesarean Delivery
Brief Title: Effects of Epidural Lidocaine on the Pharmacokinetic and Pharmacodynamic Profiles of DepoDur® After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brendan Carvalho, MD, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-07022008-1228
Record Dates: First submitted 2008-10-23; First posted 2008-12-09 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-09

CONDITIONS: Epidural Analgesia, Obstetric

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DepoDur following epidural lidocaine (Active Comparator): Epidural DepoDur was administered 60 minutes after an epidural Lidocaine top-up for surgical anesthetic in cesarean section patients.
  Interventions: Drug: DepoDur following epidural lidocaine
- DepoDur following spinal anesthetic (Active Comparator): Epidural DepoDur was administered 60 minutes after a standard spinal anesthetic. No prior epidural local anesthetic was used prior to DepoDur in this group assignment.
  Interventions: Drug: DepoDur following spinal anesthetic

INTERVENTIONS:
Drug: DepoDur following epidural lidocaine — All participant underwent cesarean delivery. An epidural "top-up" anesthetic consisting of 2% lidocaine with epinephrine 1:200,000 and sodium bicarbonate (1 meq per 10 mL lidocaine) was given. The lidocaine solution was administered in 5 mL increments every 2.5 minutes until a T6 sensory level to touch was attained. Patients also received a 100 mcg dose of fentanyl epidurally after the lidocaine solution had been administered.
  Provided delivery had occurred at least 60 minutes after the initial lidocaine administration, patients received EREM 8 mg (DepoDur™) administered through the epidural catheter. A 2 mL epidural saline flush was administered before and after drug administration.
  Other Names: DepoDur™; EREM (Extended Release Epidural Morphine)
  Arms: DepoDur following epidural lidocaine
Drug: DepoDur following spinal anesthetic — Participants underwent an elective cesarean delivery with a combined spinal/epidural. All patients received 12 mg hyperbaric bupivacaine with 20 mcg fentanyl administered intrathecally. No local anesthetic was administered through the catheter. The combined spinal-epidural was performed at the L2/L3 or L3/L4 interspace and the intrathecal dose was injected over 5-10 s. A multiple orifice epidural catheter was threaded 5 cm into the epidural space.
  Provided delivery had occurred 60 minutes after the intrathecal dose patients received EREM 8 mg (DepoDur™) through the epidural catheter. A 2 mL epidural saline flush was administered before and after drug.
  Other Names: DepoDur; EREM; extended release epidural morphine
  Arms: DepoDur following spinal anesthetic

SUMMARY:
To evaluate the levels of morphine in a patient's blood when morphine is given into the epidural space in the form of DepoDur® either alone or following a dose of lidocaine also given in the epidural space.

DETAILED DESCRIPTION:
To evaluate the levels of morphine in a patient's blood when morphine is given into the epidural space in the form of DepoDur® either alone or following a dose of lidocaine also given in the epidural space. Specifically, we are looking at pregnant women undergoing cesarean delivery who will be receiving these medications. A secondary objective is to evaluate how well DepoDur® works for pain control, as well as its safety, when it is given either alone or following a dose of epidural lidocaine.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will include healthy parturients between the ages of 18 and 40 who have American Society of Anesthesiologists physical status I or II, have an uncomplicated, singleton, term pregnancy, and are scheduled to undergo cesarean delivery.

Exclusion Criteria:

Exclusion criteria for the study will included refusal to participate, American Society of Anesthesiologists physical status III or higher or any severe uncontrolled medical condition, significant systemic medical or obstetric disease, morbid obesity, opioid, Nonsteroidal Antiinflammatory Drug (NSAID), or local anesthetic allergy or intolerance, chronic analgesic or antidepressant use, accidental dural puncture, ineffective spinal or epidural, and conversion to general anesthesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 patients enrolled at Stanford clinics
Pre-assignment Details: The patients were divided into 2 groups: group E (epidural) consisted of patients undergoing elective cesarean delivery or undergoing nonelective cesarean delivery during labor. Group SE (Spinal-Epidural) consisted of patients undergoing an elective cesarean delivery. Patients received an anesthetic consisting of a combined spinal-epidural.
Groups:
- Epidural DepoDur Following Epidural Lidocaine Administration: Epidural DepoDur was administered 60 minutes after an epidural Lidocaine top-up for surgical anesthetic in cesarean section patients.
- Epidural DepoDur Following Spinal Anesthetic: Epidural DepoDur was administered 60 minutes after a standard spinal anesthetic. No prior epidural local anesthetic was used prior to DepoDur in this group assignment.
Period: Overall Study
Arm/Group | Epidural DepoDur Following Epidural Lidocaine Administration | Epidural DepoDur Following Spinal Anesthetic
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Epidural DepoDur Following Epidural Lidocaine Administration: Epidural DepoDur was administered 60 minutes after an epidural Lidocaine top-up for surgical anesthetic in cesarean section patients.
  DepoDur: All participant underwent cesarean delivery. An epidural "top-up" anesthetic consisting of 2% lidocaine with epinephrine 1:200,000 and sodium bicarbonate (1 meq per 10 mL lidocaine) was given. The lidocaine solution was administered in 5 mL increments every 2.5 minutes until a T6 sensory level to touch was attained. Patients also received a 100 mcg dose of fentanyl epidurally after the lidocaine solution had been administered.
  Provided delivery had occurred at least 60 minutes after the initial lidocaine administration, patients received EREM 8 mg (DepoDur™) administered through the epidural catheter. A 2 mL epidural saline flush was administered before and after drug administration.
- Epidural DepoDur Following Spinal Anesthetic: Epidural DepoDur was administered 60 minutes after a standard spinal anesthetic. No prior epidural local anesthetic was used prior to DepoDur in this group assignment.
  DepoDur: Participants underwent an elective cesarean delivery with a combined spinal/epidural. All patients received 12 mg hyperbaric bupivacaine with 20 mcg fentanyl administered intrathecally. No local anesthetic was administered through the catheter. The combined spinal-epidural was performed at the L2/L3 or L3/L4 interspace and the intrathecal dose was injected over 5-10 s. A multiple orifice epidural catheter was threaded 5 cm into the epidural space.
  Provided delivery had occurred 60 minutes after the intrathecal dose patients received EREM 8 mg (DepoDur™) through the epidural catheter. A 2 mL epidural saline flush was administered before and after drug.
- Total: Total of all reporting groups
Arm/Group | Epidural DepoDur Following Epidural Lidocaine Administration | Epidural DepoDur Following Spinal Anesthetic | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (5) | 36 (3) | 34 (4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Extended Release Epidural Morphine (EREM)
Description: The primary end point was to evaluate the pharmacokinetic profiles of EREM after either no epidural lidocaine or after an epidural lidocaine top-up for cesarean delivery.
Time Frame: a plasma sample at 0, 5, 10, 15, and 30 minutes, and 1, 4, 8, 12, 24, 36, 48, and 72 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Epidural DepoDur Following Epidural Lidocaine Administration | Epidural DepoDur Following Spinal Anesthetic
Number analyzed (Participants) | 15 | 14
ng/mL | 11.1 (4.9) | 8.3 (7.1)

ADVERSE EVENTS:
Description: Serious adverse events were not collected. None were anticipated.
Arm/Group | Epidural DepoDur Following Epidural Lidocaine Administration | Epidural DepoDur Following Spinal Anesthetic
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 11/15 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural DepoDur Following Epidural Lidocaine Administration (N=15) | Epidural DepoDur Following Spinal Anesthetic (N=14)
hypotension ( 25% reduction in systolic blood pressure from baseline) (Vascular disorders) | 0 (0) | 1 (1)
supplemental oxygen (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
oxygen desaturations (defined as oxygen saturations 93%) (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No